





Initiale

Study to measure the change in heart rate when blowing in to a device, which gives resistance to exhalation (Valsalva Manoeuvre).

## ETHICS REFERENCE NUMBER: 17/06/127

## CONSENT FORM FOR PARTICIPANTS VERSION NUMBER: 4.1 01/11/17

I have read the Information Sheet Version Number 4.1 Dated 01/11/17 concerning this project and understand what it is about. All my questions have been answered to my satisfaction. I understand that I am free to request further information at any stage. I know that:

| | rinted name of researcher) his project has been reviewed and Rese | (Signature of researcher) approved by the University of Earch Ethics Committees | (Date)<br>Exeter Medical School |
|---|---|---|---|
| (Printed name of participant) (Signature of participant) | | (Date) | |
| I agree to take part in this project. | | | |
| 7. | I consent to my GP being informed in the unlikely event that an unexpected abnormality is identified during the study. | | |
| 6. | I understand that anonymous data collected during the study may<br>be looked at by individuals from the Research Team, from<br>regulatory authorities or from the NHS Trust, where it is relevant to<br>my taking part in this research. I give permission for these<br>individuals to have access to my records. | | |
| 5. | The results of the project may be purpreserved. | | |
| 4. | Data will be retained for up to 5 yea consent for its use in related studies | | |
| 3. | All data collected during the study will be retained in secure storage; | | |
| 2. | I am free to withdraw from the p disadvantage; | | |
| 1. | My participation in the project is entirely voluntary; | | |

1

UEMS REC V4.1 Nov 2017